CLINICAL TRIAL: NCT05321186
Title: Minimally Invasive Surgical Management of Traumatic Spinopelvic Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelazim Abdelrahim Hassan, Assistant Lecturer of Orthopedics and Trauma Surgery, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Spinopelvic instability
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: SPINAL Fracture
Keywords: spinopelvic instability; spinoplevic dissociation; spinopelvic fixation; lumbopelvic fixation
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Intervention Model Description: the study will be a prospective interventional case series.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- minimally invasive spinopelvic fixation. (Other): the arm will include skeletally mature patients (between the age of 18-60) presenting with sacral fractures (provided that the fracture line passes below the level of S2) associated with lumbosacral instability) with the following inclusion and exclusion criteria.
  1. Inclusion criteria:
     1. Unilateral or bilateral L5-S1 facet fractures (AO classification type C1 and C2)
     2. Spinopelvic dissociation (AO type C3)
     3. Traumatic lumbosacral dislocation
  2. Exclusion criteria:
     1. unwillingness to participate in the study
     2. pathological fractures
     3. other medical comorbidities that preclude surgical intervention.
  Interventions: Procedure: minimally invasive spinopelvic fixation

INTERVENTIONS:
Procedure: minimally invasive spinopelvic fixation — Bilateral percutaneous L4 and L5 pedicle screws will be placed under fluoroscopic guidance with Jamshidi needles, and these were will also be used the iliac fixation via percutaneous S2 alar iliac screws.
  Cases presenting with significant instability, minimally invasive Transforaminal lumbar interbody fusion (MIS-TLIF) will be performed. Additionally, in cases with neurological deficit, posterior decompression will be performed.

SUMMARY:
the main aim of this study is to evaluate the results of performing minimally invasive surgical management for cases with traumatic spinopelvic instability and spinopelvic dissociation. This will include using percutaneous pedicle and S2 alar iliac screws, minimally invasive transforaminal lumbar interbody fusion and transtubular posterior decompression.

DETAILED DESCRIPTION:
Study Procedure:

1. Patient enrollment and pre-operative evaluation:

   Upon Arrival, the patient will be managed in the emergency department according to the Advanced Trauma Life Support (ATLS) protocol. After achieving the haemodynamic stability, in cases of shock, X-rays (AP and lateral view of the lumbosacral region, inlet and outlet views of the pelvis) and CT scan of the pelvis will be performed. If the fracture pattern fits the inclusion criteria, the patient will be offered to enroll in the study and the patient will be prepared for surgery.
2. Surgery:

   The surgery will be performed under general anaesthesia and fluoroscopic guidance. The patients will be positioned prone on an open top of a radiolucent table with large bumps under the thighs to accentuate an extension force on the legs which will be the main reduction maneuver in the surgical procedure.

   Bilateral percutaneous L4 and L5 pedicle screws will be placed under fluoroscopic guidance with Jamshidi needles, and these were will also be used the iliac fixation via percutaneous S2 alar iliac screws.

   Cases presenting with significant instability, minimally invasive Transforaminal lumbar interbody fusion (MIS-TLIF) will be performed. Additionally, in cases with neurological deficit, posterior decompression will be performed.
3. Follow-up The patient will have four follow up visits (one and half month, 3month, 6month and 1 year) besides the discharge visit, during which the functional outcome scores will be filled out.

AP and lateral view pelvis x-rays will be performed every visit. CT scan, AP and lateral scanograms will be only performed on the 1-year visit.

ELIGIBILITY:
Inclusion Criteria:

Skeletally mature patients presenting with sacral fractures (provided that the fracture line passes below the level of S2) associated with lumbosacral instability showing one of the following:

1. Unilateral or bilateral L5-S1 facet fractures (AO classification type C1 and C2)
2. Spinopelvic dissociation (AO type C3)
3. Traumatic lumbosacral dislocation

Exclusion Criteria:

1. unwillingness to participate in the study
2. pathological fractures
3. other medical comorbidities that preclude surgical intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Majeed pelvic score | it will be assessed at one and half month, three month, six month and one year after the surgery
  it is a patient reported outcome score used for functional assessment after pelvic fractures.The score ranges from 0 to 100 with 0 representing the most disability and 100 the best function.

SECONDARY OUTCOMES:
Short Form 12 (SF-12) score | it will be assessed at one and half month, three month, six month and one year after the surgery
  it is a 12-item, patient-reported survey of patient health.The score ranges from 0 to 100, with higher scores indicating better physical and mental health functioning.
Oswestry disability index (ODI): | it will be assessed at one and half month, three month, six month and one year after the surgery
  it is a Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain.
Visual analogue scale of pain (VAS) | it will be assessed at one and half month, three month, six month and one year after the surgery
  It is a patient reported tool for assessment of pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.
AO PROST | it will be assessed at one and half month, three month, six month and one year after the surgery
  it is a specific patient reported outcome score designed for spine trauma patients.It consists of 19 questions on a broad range of aspects of functioning on a 0-100 numeric rating scale with 0 indicating no function at all and 100 the pre-injury level of function.
lumbar lordosis | it will be assessed at one and half month, three month, six month and one year after the surgery
  it will measured in degrees on plain standing lateral lumbosacral x-rays.
Gibbons' criteria | it will be assessed at one and half month, three month, six month and one year after the surgery
  it is a classification used to stratify patients with neurological deficit associated with pelvic injuries
pelvic incidence | it will be assessed at one and half month, three month, six month and one year after the surgery
  it will be measured in degrees on plain standing lateral lumbosacral x-rays.
AP translation | it will be assessed at one and half month, three month, six month and one year after the surgery
  it will be measured in millimetres on inlet and outlet pelvic x-rays.
vertical translation | it will be assessed at one and half month, three month, six month and one year after the surgery
  it will be measured in millimetres on plain standing AP pelvic x-rays.
sacral table angle | it will be assessed at one and half month, three month, six month and one year after the surgery
  it will be measured in degrees on plain standing lateral lumbosacral x-rays.
sacral kyphosis angle | it will be assessed at one and half month, three month, six month and one year after the surgery
  it will be measured in degrees on plain standing lateral lumbosacral x-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A A Hassan, MBBCh, MSc, Principal Investigator — Assistant Lecturer, Faculty of Medicine, Assiut University

IPD SHARING:
Plan to Share IPD: No